CLINICAL TRIAL: NCT01612338
Title: Interventions to Increase Screening Utilization by Breast Cancer Survivors and Their High Risk Female Relatives: Using Cancer Surveillance and the Michigan Genomics Academic-Practice Partnership
Brief Title: Interventions to Increase Screening by Breast Cancer Survivors and Their High Risk Female Relatives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Michigan Department of Community Health (Other)
Responsible Party: Principal Investigator, Maria Katapodi, PhD, RN, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 5U48DP001901-03 (NIH)
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2014-10

CONDITIONS: Breast Cancer; Breast Cancer in Young Women; Breast Cancer in Women With a Strong Family History
Keywords: breast cancer; young age of onset; family history; screening interventions; family support
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Targeted (Experimental): Targeted letter and booklet
  Interventions: Behavioral: Targeted
- Tailored (Experimental): Tailored letter and booklet, enhanced family communication and support brochure
  Interventions: Behavioral: Enhanced Tailored

INTERVENTIONS:
Behavioral: Targeted — Targeted letter and booklet
  Arms: Targeted
Behavioral: Enhanced Tailored — Tailored letter and booklet, enhanced family communication and support brochure
  Arms: Tailored

SUMMARY:
The University of Michigan (UM) Schools of Nursing, Public Health, and Medicine, the Michigan Department of Community Health (MDCH) and the Michigan Cancer Consortium (MCC) are conducting a multidisciplinary academic/practice three-year project to increase appropriate breast cancer screening for young breast cancer survivors and their cancer-free, female relatives at greatest risk for breast cancer. The aims of this project are to: 1) identify and survey 3000 breast cancer survivors reported to the Michigan Cancer Surveillance Program who were diagnosed between the ages of 20-45 years regarding their breast cancer screening utilization; 2) identify and survey the survivors' female relatives regarding their breast cancer screening utilization; and 3) implement two versions (targeted vs. enhanced tailored) of an evidence-based intervention recommended by the Guide to Community Preventive Services to increase breast cancer screening. A follow-up survey will assess the effectiveness of each intervention on a) breast cancer screening utilization; b) perceived barriers and facilitators to screening; c) self-efficacy in utilizing screening services; d) family support related to screening; e) knowledge of the genetics of breast cancer and personal risk factors; and f) satisfaction with the intervention.

DETAILED DESCRIPTION:
The University of Michigan (UM) Schools of Nursing, Public Health, and Medicine, the Michigan Department of Community Health (MDCH) and the Michigan Cancer Consortium (MCC) propose a multidisciplinary academic/practice three-year project to increase appropriate breast cancer screening utilization for young breast cancer survivors (YBCS), and their cancer-free, female relatives at greatest risk for breast cancer (high-risk relatives). The aims of this project are to: 1) identify and survey 3000 breast cancer survivors reported to the Michigan Cancer Surveillance Program who were diagnosed between the ages of 25-45 years regarding their breast cancer screening utilization; 2) identify and survey YBCS' high-risk relatives regarding their breast cancer screening utilization; and 3) implement two versions (targeted vs. enhanced tailored) of an evidence-based intervention recommended by the Guide to Community Preventive Services to increase breast cancer screening. Aim 1, will be accomplished in year 1 by MDCH, UM and MCSP. Following approval by appropriate review boards (MDCH, UM, and MCSP), reporting facilities and physicians of record, 3000 YBCS will be mailed a request to participate in the project and a baseline survey. The baseline survey will obtain information on the YBCS's: a) willingness to participate; b) current breast cancer screening utilization; c) perceived barriers and facilitators to screening and other outcomes related to breast cancer screening; d) identification of high-risk relatives to participate in the study and interest in serving as an advocate for their high-risk relatives to participate. Aim 2, will be accomplished in year 2 by the UM and MDCH. Based on the information provided by YBCS, the MDCH will identify up to two high-risk relatives per YBCS. UM and MDCH will mail YBCS who agree to participate in the study baseline surveys to distribute to their selected high-risk relatives. The baseline survey to high-risk relatives will obtain information on their: a) willingness to participate in the project; b) current breast cancer screening utilization; and c) perceived barriers and facilitators to screening and other outcomes related to breast cancer screening. Aim 3, will be accomplished by UM and MDCH. YBCS and their high-risk relatives will be randomized (as a family unit) to receive two versions of a small media, evidence-based intervention aiming to increase appropriate utilization of breast cancer screening services and other outcomes. In year 2-3, 9 months after YBCS and high-risk female relatives receive the intervention, UM will mail a follow-up survey to YBCS and their high-risk relatives to evaluate the effectiveness of each intervention version on: a) breast cancer screening utilization; b) perceived barriers and facilitators to screening; c) self-efficacy in utilizing screening services; d) family support related to screening; e) knowledge of the genetics of breast cancer and personal risk factors; and f) satisfaction with the intervention. The State of Michigan is considered a national leader in cancer prevention, control, and public health genomics. Key partners have significant prior experience in conducting studies with cancer survivors and their high-risk relatives. This project would greatly enhance state efforts in cancer prevention and control.

ELIGIBILITY:
Inclusion Criteria:

* For breast cancer survivors

  * Female
  * 20-64 years of age
  * Being diagnosed with invasive breast cancer between 20 and 45 years of age
  * Being diagnosed with DCIS between 20 and 45 years of age
  * Michigan resident at time of diagnosis
  * able to read and understand English
  * not currently pregnant, incarcerated, or institutionalized
* For high risk relatives

  * Female
  * First- or second- degree relatives of survivor
  * 25-64 years of age
  * US resident
  * Able to read and understand English
  * Unaffected with any type of cancer
  * Not currently pregnant, incarcerated, or institutionalized
  * Survivor is willing to contact

Exclusion Criteria:

-

Ages: 20 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1290 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
breast cancer screening | 9 months
  self report of mammogram and clinical breast exam
genetic counseling | 9 months
  self report of obtaining genetic counseling

SECONDARY OUTCOMES:
barriers to screening | 9 months
  Barriers and Facilitators to Mammography
knowledge of breast cancer genetics | 9 months
  Genetic literacy

CONTACTS AND LOCATIONS:
Overall Officials: Maria C. Katapodi, PhD, Principal Investigator — University of Michigan School of Nursing
Locations (2):
- United States (2):
  - University of Michigan School of Nursing, Ann Arbor, Michigan
  - Michigan Department of Community Health, Lansing, Michigan

REFERENCES:
- [Background] Katapodi MC, Northouse LL, Schafenacker AM, Duquette D, Duffy SA, Ronis DL, Anderson B, Janz NK, McLosky J, Milliron KJ, Merajver SD, Duong LM, Copeland G. Using a state cancer registry to recruit young breast cancer survivors and high-risk relatives: protocol of a randomized trial testing the efficacy of a targeted versus a tailored intervention to increase breast cancer screening. BMC Cancer. 2013 Mar 1;13:97. doi: 10.1186/1471-2407-13-97. PMID 23448100
- [Result] Jones T, Lockhart JS, Mendelsohn-Victor KE, Duquette D, Northouse LL, Duffy SA, Donley R, Merajver SD, Milliron KJ, Roberts JS, Katapodi MC. Use of Cancer Genetics Services in African-American Young Breast Cancer Survivors. Am J Prev Med. 2016 Oct;51(4):427-36. doi: 10.1016/j.amepre.2016.03.016. Epub 2016 Apr 23. PMID 27117712
- [Result] Katapodi MC, Duquette D, Yang JJ, Mendelsohn-Victor K, Anderson B, Nikolaidis C, Mancewicz E, Northouse LL, Duffy S, Ronis D, Milliron KJ, Probst-Herbst N, Merajver SD, Janz NK, Copeland G, Roberts S. Recruiting families at risk for hereditary breast and ovarian cancer from a statewide cancer registry: a methodological study. Cancer Causes Control. 2017 Mar;28(3):191-201. doi: 10.1007/s10552-017-0858-2. Epub 2017 Feb 14. PMID 28197806
- [Result] Jones T, Duquette D, Underhill M, Ming C, Mendelsohn-Victor KE, Anderson B, Milliron KJ, Copeland G, Janz NK, Northouse LL, Duffy SM, Merajver SD, Katapodi MC. Surveillance for cancer recurrence in long-term young breast cancer survivors randomly selected from a statewide cancer registry. Breast Cancer Res Treat. 2018 May;169(1):141-152. doi: 10.1007/s10549-018-4674-5. Epub 2018 Jan 20. PMID 29353367
- [Result] Katapodi MC, Ellis KR, Schmidt F, Nikolaidis C, Northouse LL. Predictors and interdependence of family support in a random sample of long-term young breast cancer survivors and their biological relatives. Cancer Med. 2018 Oct;7(10):4980-4992. doi: 10.1002/cam4.1766. Epub 2018 Sep 5. PMID 30187678
- [Result] Nikolaidis C, Duquette D, Mendelsohn-Victor KE, Anderson B, Copeland G, Milliron KJ, Merajver SD, Janz NK, Northouse LL, Duffy SA, Katapodi MC. Disparities in genetic services utilization in a random sample of young breast cancer survivors. Genet Med. 2019 Jun;21(6):1363-1370. doi: 10.1038/s41436-018-0349-1. Epub 2018 Nov 2. PMID 30385886
- [Derived] Ellis KR, Koechlin H, Rudaz M, Gerido LH, Hecht HK, Jones C, Raji D, Northouse L, Katapodi M. Predictors and Interdependence of Quality of Life in a Random Sample of Long-Term Young Breast Cancer Survivors and Their Biological Relatives. Cancer Med. 2024 Oct;13(20):e70328. doi: 10.1002/cam4.70328. PMID 39470180